CLINICAL TRIAL: NCT06521879
Title: Improved Gastrointestinal Tolerance and Iron Status Via Probiotic Use in Iron Deficiency Anemia Patients Initiating Oral Iron Replacement
Brief Title: Probiotic Use in Oral Iron Replacement Deficiency Anemia Patients Initiating Oral Iron Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-265
Record Dates: First submitted 2024-07-14; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Iron Deficiency Anemia Treatment; Iron Deficiency Anemia
Keywords: iron deficiency anemia; oral iron replacement; probiotic supplementation; Lactobacillus plantarum 299v; gastrointestinal tolerability; iron status markers
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned via simple randomization method (computer- generated random number sequence)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IRT-Only (No Intervention): Iron deficiency anemia patients receive iron replacement therapy alone.
- IRT-Pro (Experimental): Iron deficiency anemia patients receive iron replacement therapy plus L. plantarum 299v probiotic support
  Interventions: Dietary Supplement: Lactobacillus plantarum 299v probiotic support

INTERVENTIONS:
Dietary Supplement: Lactobacillus plantarum 299v probiotic support — Addition of Lactobacillus plantarum 299v (L. plantarum 299v) probiotic supplementation to iron replacement therapy.
  Arms: IRT-Pro

SUMMARY:
Investigation of gastrointestinal tolerability, treatment compliance and iron status markers in patients with iron deficiency anemia who received oral iron replacement therapy with versus without concomitant probiotic supplementation

DETAILED DESCRIPTION:
A total of 295 patients, with newly diagnosed iron deficiency anemia (IDA) who were planned to receive routine oral IRT were included in this prospective randomized non-placebo, controlled 3-month follow-up study. Patients were randomly assigned via simple randomization method to receive either iron replacement therapy (IRT) alone or IRT plus L. plantarum 299v probiotic support . Adult (aged older than18 years) treatment-naïve patients diagnosed with newly diagnosed IDA without previous IRT were included in the study, while those with irritable bowel syndrome, previous IRT therapy or intolerance to IRT and those with a known chronic disease (i.e., inflammatory bowel disease (IBD), celiac disease) or untreated active menometrorrhagia and hemorrhoid were excluded from the study.

All patients received IRT with ferrous sulfate (Fe2 + ) preparation (100 mg, once daily) for 3 months, while those in the IRT-Pro group also received daily (10B CFU) L. plantarum 299v probiotic supplementation for 30 days starting from the first day of IRT.

Data on gastrointestinal intolerance symptoms (loss of appetite, nausea, vomiting, abdominal pain, diarrhea, constipation and bloating) were recorded at three time points including baseline, within the first 30 days of IRT and at any time during 3-month IRT.

Serum hemoglobin levels (g/dL) and serum iron status markers including ferritin (ng/mL), iron (µg/dL), total iron binding capacity (TIBC, µg/dL) and transferrin saturation (%) were recorded at baseline and at 3 rd month of IRT. Data on treatment discontinuation were also recorded in study groups along with comparison of study variables in patients with vs. without treatment discontinuation within the first 30 days of IRT.

At least 189 patients were calculated to be included via sample size estimation (G*Power 3.1.9 program) based on a power of 80 % at a type I error of 0.05, and an effect size (w=0.261) calculated using data from a previous study by Cekin et al. .

Given the high likelihood of missing data, a total of 200 patients were planned to be included in the study population with the use of 25% lost to follow up ratio. Statistical analysis was made using IBM SPSS Statistics for Windows, Version 22.0 (IBM Corp., Armonk, NY). Pearson chi-square test, Fisher's exact test and Mc-Nemar test were used for analysis of categorical variables. Mann-Whitney U test was used for analysis of non-normally distributed numerical data while independent sample t test was used for normally distributed data. The number needed to treat (NNT) analysis was performed to determine how many patients must receive IRT-Pro instead of IRT per se to prevent one additional treatment discontinuation. Data are expressed as mean ± standard deviation (SD), median, inter-quartile range (IQR), minimum-maximum and percent (%) where appropriate. p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naïve patients diagnosed with newly diagnosed iron deficiency anemia

Exclusion Criteria:

* Irritable bowel syndrome
* Celiac disease
* Untreated active menometrorrhagia
* Hemorrhoidal disease
* Previous iron replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 295 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Tolerance and Treatment Compliance in Iron Deficiency Anemia Patients Using Oral Iron with or without Lactobacillus plantarum 299v Probiotic Supplementation | 3 months
  To investigate gastrointestinal tolerability and treatment compliance in patients with iron deficiency anemia who received oral iron replacement therapy with versus without concomitant Lactobacillus plantarum 299v (L. plantarum 299v) probiotic supplementation. Gastrointestinal intolerance symptoms (loss of appetite, nausea, vomiting, abdominal pain, diarrhea, constipation, and bloating) will be assessed using a structured questionnaire with yes or no questions.
  Measurement Tool: Structured Questionnaire
  Data Collection Points: Baseline, within the first 30 days of iron replacement therapy (IRT), and at any time during the 3-month IRT.
  Scale Description: The questionnaire will include yes or no questions to determine the presence of gastrointestinal intolerance symptoms. A "yes" response indicates the presence of a symptom, and a "no" response indicates its absence.

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Koker, MD, Principal Investigator — Antalya Training and Research Hospital; Yasin Sahinturk, MD, Study Chair — Antalya Training and Research Hospital; Gulhan Ozcelik Koker, MD, Study Chair — Antalya Training and Research Hospital; Ali Coskuner, MD, Study Chair — Antalya Training and Research Hospital; Merve Eren Durmuş, MD, Study Chair — Antalya Training and Research Hospital; Mutlu M Catli, MD, Study Chair — Antalya Training and Research Hospital; Ayhan H Cekin, MD, Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stevens GA, Finucane MM, De-Regil LM, Paciorek CJ, Flaxman SR, Branca F, Pena-Rosas JP, Bhutta ZA, Ezzati M; Nutrition Impact Model Study Group (Anaemia). Global, regional, and national trends in haemoglobin concentration and prevalence of total and severe anaemia in children and pregnant and non-pregnant women for 1995-2011: a systematic analysis of population-representative data. Lancet Glob Health. 2013 Jul;1(1):e16-25. doi: 10.1016/S2214-109X(13)70001-9. Epub 2013 Jun 25. PMID 25103581
- [Background] Kumar SB, Arnipalli SR, Mehta P, Carrau S, Ziouzenkova O. Iron Deficiency Anemia: Efficacy and Limitations of Nutritional and Comprehensive Mitigation Strategies. Nutrients. 2022 Jul 20;14(14):2976. doi: 10.3390/nu14142976. PMID 35889932
- [Background] Seo H, Yoon SY, Ul-Haq A, Jo S, Kim S, Rahim MA, Park HA, Ghorbanian F, Kim MJ, Lee MY, Kim KH, Lee N, Won JH, Song HY. The Effects of Iron Deficiency on the Gut Microbiota in Women of Childbearing Age. Nutrients. 2023 Jan 30;15(3):691. doi: 10.3390/nu15030691. PMID 36771397
- [Background] Zakrzewska Z, Zawartka A, Schab M, Martyniak A, Skoczen S, Tomasik PJ, Wedrychowicz A. Prebiotics, Probiotics, and Postbiotics in the Prevention and Treatment of Anemia. Microorganisms. 2022 Jun 30;10(7):1330. doi: 10.3390/microorganisms10071330. PMID 35889049
- [Background] Goodnough LT, Nemeth E, Ganz T. Detection, evaluation, and management of iron-restricted erythropoiesis. Blood. 2010 Dec 2;116(23):4754-61. doi: 10.1182/blood-2010-05-286260. Epub 2010 Sep 8. PMID 20826717
- [Background] Vonderheid SC, Tussing-Humphreys L, Park C, Pauls H, OjiNjideka Hemphill N, LaBomascus B, McLeod A, Koenig MD. A Systematic Review and Meta-Analysis on the Effects of Probiotic Species on Iron Absorption and Iron Status. Nutrients. 2019 Dec 3;11(12):2938. doi: 10.3390/nu11122938. PMID 31816981
- [Background] Korcok DJ, Trsic-Milanovic NA, Ivanovic ND, Dordevic BI. Development of Probiotic Formulation for the Treatment of Iron Deficiency Anemia. Chem Pharm Bull (Tokyo). 2018 Apr 1;66(4):347-352. doi: 10.1248/cpb.c17-00634. Epub 2018 Jan 19. PMID 29353864
- [Background] Rusu IG, Suharoschi R, Vodnar DC, Pop CR, Socaci SA, Vulturar R, Istrati M, Morosan I, Farcas AC, Kerezsi AD, Muresan CI, Pop OL. Iron Supplementation Influence on the Gut Microbiota and Probiotic Intake Effect in Iron Deficiency-A Literature-Based Review. Nutrients. 2020 Jul 4;12(7):1993. doi: 10.3390/nu12071993. PMID 32635533
- [Background] Bazeley JW, Wish JB. Recent and Emerging Therapies for Iron Deficiency in Anemia of CKD: A Review. Am J Kidney Dis. 2022 Jun;79(6):868-876. doi: 10.1053/j.ajkd.2021.09.017. Epub 2021 Nov 7. PMID 34758368
- [Background] Kumar A, Sharma E, Marley A, Samaan MA, Brookes MJ. Iron deficiency anaemia: pathophysiology, assessment, practical management. BMJ Open Gastroenterol. 2022 Jan;9(1):e000759. doi: 10.1136/bmjgast-2021-000759. PMID 34996762
- [Background] Gomez-Ramirez S, Brilli E, Tarantino G, Munoz M. Sucrosomial(R) Iron: A New Generation Iron for Improving Oral Supplementation. Pharmaceuticals (Basel). 2018 Oct 4;11(4):97. doi: 10.3390/ph11040097. PMID 30287781
- [Background] Auerbach M, Adamson JW. How we diagnose and treat iron deficiency anemia. Am J Hematol. 2016 Jan;91(1):31-8. doi: 10.1002/ajh.24201. Epub 2015 Nov 17. PMID 26408108
- [Background] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159
- [Background] Deschemin JC, Noordine ML, Remot A, Willemetz A, Afif C, Canonne-Hergaux F, Langella P, Karim Z, Vaulont S, Thomas M, Nicolas G. The microbiota shifts the iron sensing of intestinal cells. FASEB J. 2016 Jan;30(1):252-61. doi: 10.1096/fj.15-276840. Epub 2015 Sep 14. PMID 26370847
- [Background] Jaeggi T, Kortman GA, Moretti D, Chassard C, Holding P, Dostal A, Boekhorst J, Timmerman HM, Swinkels DW, Tjalsma H, Njenga J, Mwangi A, Kvalsvig J, Lacroix C, Zimmermann MB. Iron fortification adversely affects the gut microbiome, increases pathogen abundance and induces intestinal inflammation in Kenyan infants. Gut. 2015 May;64(5):731-42. doi: 10.1136/gutjnl-2014-307720. Epub 2014 Aug 20. PMID 25143342
- [Background] Hoppe M, Onning G, Berggren A, Hulthen L. Probiotic strain Lactobacillus plantarum 299v increases iron absorption from an iron-supplemented fruit drink: a double-isotope cross-over single-blind study in women of reproductive age. Br J Nutr. 2015 Oct 28;114(8):1195-202. doi: 10.1017/S000711451500241X. PMID 26428277
- [Background] Wells JM. Immunomodulatory mechanisms of lactobacilli. Microb Cell Fact. 2011 Aug 30;10 Suppl 1(Suppl 1):S17. doi: 10.1186/1475-2859-10-S1-S17. Epub 2011 Aug 30. PMID 21995674
- [Background] Goossens D, Jonkers D, Russel M, Thijs A, van den Bogaard A, Stobberingh E, Stockbrugger R. Survival of the probiotic, L. plantarum 299v and its effects on the faecal bacterial flora, with and without gastric acid inhibition. Dig Liver Dis. 2005 Jan;37(1):44-50. doi: 10.1016/j.dld.2004.07.018. PMID 15702859
- [Background] Ducrotte P, Sawant P, Jayanthi V. Clinical trial: Lactobacillus plantarum 299v (DSM 9843) improves symptoms of irritable bowel syndrome. World J Gastroenterol. 2012 Aug 14;18(30):4012-8. doi: 10.3748/wjg.v18.i30.4012. PMID 22912552
- [Background] Niedzielin K, Kordecki H, Birkenfeld B. A controlled, double-blind, randomized study on the efficacy of Lactobacillus plantarum 299V in patients with irritable bowel syndrome. Eur J Gastroenterol Hepatol. 2001 Oct;13(10):1143-7. doi: 10.1097/00042737-200110000-00004. PMID 11711768
- [Background] Bering S, Sjoltov L, Wrisberg SS, Berggren A, Alenfall J, Jensen M, Hojgaard L, Tetens I, Bukhave K. Viable, lyophilized lactobacilli do not increase iron absorption from a lactic acid-fermented meal in healthy young women, and no iron absorption occurs in the distal intestine. Br J Nutr. 2007 Nov;98(5):991-7. doi: 10.1017/S0007114507761809. Epub 2007 Sep 3. PMID 17764597
- [Background] Scheers N, Rossander-Hulthen L, Torsdottir I, Sandberg AS. Increased iron bioavailability from lactic-fermented vegetables is likely an effect of promoting the formation of ferric iron (Fe(3+)). Eur J Nutr. 2016 Feb;55(1):373-82. doi: 10.1007/s00394-015-0857-6. Epub 2015 Feb 12. PMID 25672527
- [Background] Sahin K, Sahinturk Y, Koker G, Ozcelik Koker G, Bostan F, Kok M, Uyar S, Cekin AH. Metformin with Versus without Concomitant Probiotic Therapy in Newly Diagnosed Patients with Type 2 Diabetes or Prediabetes: A Comparative Analysis in Relation to Glycemic Control, Gastrointestinal Side Effects, and Treatment Compliance. Turk J Gastroenterol. 2022 Nov;33(11):925-933. doi: 10.5152/tjg.2022.211063. PMID 36098362
- [Background] Cekin AH, Sahinturk Y, Akbay Harmandar F, Uyar S, Yolcular BO, Cekin Y. Use of probiotics as an adjuvant to sequential H. pylori eradication therapy: impact on eradication rates, treatment resistance, treatment-related side effects, and patient compliance. Turk J Gastroenterol. 2017 Jan;28(1):3-11. doi: 10.5152/tjg.2016.0278. Epub 2016 Dec 23. PMID 28007678
- [Background] Endo H, Higurashi T, Hosono K, Sakai E, Sekino Y, Iida H, Sakamoto Y, Koide T, Takahashi H, Yoneda M, Tokoro C, Inamori M, Abe Y, Nakajima A. Efficacy of Lactobacillus casei treatment on small bowel injury in chronic low-dose aspirin users: a pilot randomized controlled study. J Gastroenterol. 2011 Jul;46(7):894-905. doi: 10.1007/s00535-011-0410-1. Epub 2011 May 10. PMID 21556830
- [Background] Axling U, Onning G, Martinsson Niskanen T, Larsson N, Hansson SR, Hulthen L. The effect of Lactiplantibacillus plantarum 299v together with a low dose of iron on iron status in healthy pregnant women: A randomized clinical trial. Acta Obstet Gynecol Scand. 2021 Sep;100(9):1602-1610. doi: 10.1111/aogs.14153. Epub 2021 Apr 21. PMID 33880752
- [Background] OjiNjideka Hemphill N, Pezley L, Steffen A, Elam G, Kominiarek MA, Odoms-Young A, Kessee N, Hamm A, Tussing-Humphreys L, Koenig MD. Feasibility Study of Lactobacillus Plantarum 299v Probiotic Supplementation in an Urban Academic Facility among Diverse Pregnant Individuals. Nutrients. 2023 Feb 9;15(4):875. doi: 10.3390/nu15040875. PMID 36839232
- [Background] Sandberg AS, Onning G, Engstrom N, Scheers N. Iron Supplements Containing Lactobacillus plantarum 299v Increase Ferric Iron and Up-regulate the Ferric Reductase DCYTB in Human Caco-2/HT29 MTX Co-Cultures. Nutrients. 2018 Dec 8;10(12):1949. doi: 10.3390/nu10121949. PMID 30544799
- [Background] Jaramillo A, Briones L, Andrews M, Arredondo M, Olivares M, Brito A, Pizarro F. Effect of phytic acid, tannic acid and pectin on fasting iron bioavailability both in the presence and absence of calcium. J Trace Elem Med Biol. 2015 Apr;30:112-7. doi: 10.1016/j.jtemb.2014.11.005. Epub 2014 Nov 27. PMID 25544113
- [Background] Liu H, Wu W, Luo Y. Oral and intravenous iron treatment alter the gut microbiome differentially in dialysis patients. Int Urol Nephrol. 2023 Mar;55(3):759-767. doi: 10.1007/s11255-022-03377-0. Epub 2022 Sep 27. PMID 36166104
- [Background] Kujawa-Szewieczek A, Adamczak M, Kwiecien K, Dudzicz S, Gazda M, Wiecek A. The Effect of Lactobacillus plantarum 299v on the Incidence of Clostridium difficile Infection in High Risk Patients Treated with Antibiotics. Nutrients. 2015 Dec 4;7(12):10179-88. doi: 10.3390/nu7125526. PMID 26690209
- [Background] Kazmierczak-Siedlecka K, Daca A, Folwarski M, Witkowski JM, Bryl E, Makarewicz W. The role of Lactobacillus plantarum 299v in supporting treatment of selected diseases. Cent Eur J Immunol. 2020;45(4):488-493. doi: 10.5114/ceji.2020.101515. Epub 2021 Jan 25. PMID 33613097
- [Background] Serati M, Torella M. Preventing complications by persistence with iron replacement therapy: a comprehensive literature review. Curr Med Res Opin. 2019 Jun;35(6):1065-1072. doi: 10.1080/03007995.2018.1552850. Epub 2019 Jan 3. PMID 30477352
- [Background] Richards T, Breymann C, Brookes MJ, Lindgren S, Macdougall IC, McMahon LP, Munro MG, Nemeth E, Rosano GMC, Schiefke I, Weiss G. Questions and answers on iron deficiency treatment selection and the use of intravenous iron in routine clinical practice. Ann Med. 2021 Dec;53(1):274-285. doi: 10.1080/07853890.2020.1867323. PMID 33426933
- [Background] Bering S, Suchdev S, Sjoltov L, Berggren A, Tetens I, Bukhave K. A lactic acid-fermented oat gruel increases non-haem iron absorption from a phytate-rich meal in healthy women of childbearing age. Br J Nutr. 2006 Jul;96(1):80-5. doi: 10.1079/bjn20061683. PMID 16869994
- [Background] Axling U, Onning G, Combs MA, Bogale A, Hogstrom M, Svensson M. The Effect of Lactobacillus plantarum 299v on Iron Status and Physical Performance in Female Iron-Deficient Athletes: A Randomized Controlled Trial. Nutrients. 2020 Apr 30;12(5):1279. doi: 10.3390/nu12051279. PMID 32365981
- [Background] Fikri B, Ridha NR, Putri SH, Salekede SB, Juliaty A, Tanjung C, Massi N. Effects of probiotics on immunity and iron homeostasis: A mini-review. Clin Nutr ESPEN. 2022 Jun;49:24-27. doi: 10.1016/j.clnesp.2022.03.031. Epub 2022 Mar 31. PMID 35623819
- [Derived] Koker G, Sahinturk Y, Ozcelik Koker G, Coskuner MA, Eren Durmus M, Catli MM, Cekin AH. Improved gastrointestinal tolerance and iron status via probiotic use in iron deficiency anaemia patients initiating oral iron replacement: a randomised controlled trial. Br J Nutr. 2024 Nov 28;132(10):1308-1316. doi: 10.1017/S0007114524002757. Epub 2024 Nov 4. PMID 39494607